CLINICAL TRIAL: NCT01965496
Title: A Double-Blind, Multicenter, Randomized Study Evaluating the Safety, Tolerability and Pharmacokinetic/Pharmacodynamic Relationship in T2DMs Treated With 14 Weeks Injection of Polyethylene Glycol Loxenatide
Brief Title: A Phase I Study of Polyethylene Glycol Loxenatide in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: People's Liberation Army General Hospital of Chengdu Military Region (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEX168-I-05
Record Dates: First submitted 2013-06-12; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: PEX168; Phase I; titration
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — polyethylene glycol loxenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEX168 100 microgram (Experimental): PEX168 100 microgram qw sc. and the medication continued for 14 weeks
  Interventions: Drug: PEX168
- PEX168 200 microgram (Experimental): PEX168 200 microgram qw sc. and the medication start form 100 microgram qw for 4 weeks and then increased to 200 microgram qw for the 10 weeks.
  Interventions: Drug: PEX168
- PEX168 300 microgram (Experimental): PEX168 300 microgram qw sc. and the medication start form 100 microgram qw for 4 weeks and then increased to 300 microgram qw for the 10 weeks.
  Interventions: Drug: PEX168

INTERVENTIONS:
Drug: PEX168 — A injection administered subcutaneously
  Other Names: Polyethylene Glycol Loxenatide

SUMMARY:
Polyethylene Glycol Loxenatide (PEX168) is a new human glucagon-like peptide 1 (GLP-1) analogue that created on the basis of the Exenatide and modified by polyethylene glycol (PEG).

This study aims to evaluate whether the titration mode of administration could reduce the incidence of adverse reactions of PEX168, also decided to observe long-term continuous administration of PK/PD correlation.

ELIGIBILITY:
Inclusion Criteria:

1. Has been diagnosed with type 2 diabetes mellitus
2. Has been treated with either: diet and exercise alone, or with a stable regimen of one or combination of two oral antihyperglycaemic agents (except TZDs), for a minimum of 3 months prior to study start.
3. Has HbA1c of 7.5% to 11.0%, inclusive.
4. Is 20 to 72 years old, inclusive.
5. Has a body mass index (BMI) of 19 kg/m2 to 35 kg/m2, inclusive.

Exclusion Criteria:

1. Skin test of PEX168 is positive.
2. Is currently treated with any of the following excluded medications:

   * GLP-1 or GLP-1 analogues prior to study start;
   * Insulin within 6 months prior to study start;
   * Growth hormone within 6 months prior to study start;
   * Abuse of drug or alcohol within 6 months prior to study start;
   * Any clinical trials of drugs or medical instruments within 3 months prior to study start;
   * Systemic corticosteroids by oral, parenteral, or intra-articular route
   * Any drugs for weight loss or operations leading to weight instable within 2 months prior to study start;
   * Any drugs that may interfere the evaluation of safety and efficiency of investigated drugs, drugs or herbals medicine that may result in toxicity to main organs prior to study start;
3. A history or evidence of any of the following :

   * Severe hypoglycemia history (e.g., sleepiness, consciousness disorder, deliration, coma led by hypoglycemia )
   * Type 1diabetes, monogenic diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes (e.g., Cushing's syndrome or acromegaly-associated diabetes).
   * Other endocrine diseases (e.g., hyperthyreosis, hypothyroidism)
   * Acute or chronic gastrointestinal diseases that were not suitable for the trials evaluated by investigators.
   * Hypertension with SBP>140mmHg, and/or DBP >90mmHg after antihypertensive therapy.
   * Severe cardiovascular diseases histories including congestive heart failure (NYHA III or IV), unstable angina, stroke or TIA, myocardial infarction,sustained and clinically relevant ventricular arrhythmia, coronary artery bypass surgery or percutaneous coronary intervention.
   * Acute or chronic pancreatitis history, or pancreas injury history, or any high risk factors which may result in pancreatitis.
   * Malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, regardless of whether there is evidence of local recurrence or metastases.
   * Medullary thyroid carcinoma history, or multiple endocrine neoplasia history.
   * Acute metabolic complications such as ketoacidosis, lactic acidosis, or hyperosmolar state (coma) , or maculopathy , or instability of proliferative retinopathy within the past 6 months.
   * Weight change is over 10% within 3 months prior to the study start.
   * hepatitis B positive, hepatitis C antibody positive, HIV antibody positive, syphilis antibody positive.
4. Any of the following significant laboratory abnormalities:

   * Alanine aminotrasferase (ALT) and/or asparatate aminotransferase (AST)>2*upper limit of normal (ULN), and/or total bilirubin>1.5*ULN, confirmed by repeat measure;
   * Creatinine > upper limit of normal, confirmed by repeat measure, and/or proteinurea>++ and 24 hour urinary protein quantitative ≥1g.
   * Thyroid dysfunction unsuitable for this trial evaluated by investigator;
   * Hemodlastase > upper limit of normal, confirmed by repeat measure;
5. Male or female fertility are reluctant to take contraceptive method during the test, pregnancy or lactating women;
6. Any other situations which may result in the withdrawal of subjects or bring significant risk to subjects.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To assess HbA1C levels after 14 weeks continuous treatment | 14 weeks

SECONDARY OUTCOMES:
To assess Fasting blood glucose levels | 14 weeks

OTHER OUTCOMES:
To assess number of participants with Adverse Events as a Measure of Safety and Tolerability | 14 weeks
To assess the body weights after the treatment | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, M.D, Principal Investigator — People's Liberation Army General Hospital of Chengdu Military Region
Locations (1):
- People's Liberation Army General Hospital of Chengdu Military Region, Chengdu, China